CLINICAL TRIAL: NCT03446521
Title: Humoral Immune Status in Patients With Liver Cirrhosis Before and After Liver Transplantation
Brief Title: AGRA Before and After Liver Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: AGRA-TX
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: Patients undergoing liver transplantation, no intervention (study-specific) is planed
- Control Group: Respective organ donors of the included liver recipients, no intervention (study-specific) is planed

SUMMARY:
The immune system is impaired in liver cirrhotic patients, which is associated with a high risk for bacterial infections and worse outcome. A novel biomarker, acellular growth retardation ability (AGRA), can predict the development of severe infections in patients with liver cirrhosis and therefore identify patients at risk. It is still unclear, how this biomarker develops after liver transplantation and how valid its predictions are for post-operative infections. Therefore, AGRA will be measured before and after liver transplantation and predictive merit of AGRA for post-transplant infections will be tested.

DETAILED DESCRIPTION:
Cirrhosis-associated immune dysfunction syndrome (CAIDS) is a well-recognized phenomenon. It affects all immune cells as well as the humoral immune system. Because of this deficiency patients with liver cirrhosis often suffer from severe infections that can be complicated by sepsis, acute renal or liver failure, and lead to prolonged hospitalization and ultimately to the death of the patient. The humoral immune system is a first-line defence mechanism and consists of cell-free molecules that are partly produced by the liver and target pathogens through opsonisation, growth inhibition and lysis. A cirrhotic liver cannot reach its full protein expression capacity and consequently, quantitative and qualitative changes of complement factors and immunoglobulins have been observed in liver disease patients before.

Liver transplantation remains the only curative option to treat liver cirrhosis and its extrahepatic manifestations; however due to limited organ supply this option is not applicable in all cases. Therefore, liver cirrhosis and its complications (eg. infections) need to be managed by health care professionals, who often lack appropriate tools for risk assessment. To meet this clinical need, a novel biomarker was recently established (Acellular Growth Retardation Ability, short AGRA) that uses the state of the humoral immune system to predict the future occurrence of severe infection in liver disease patients. However, it is still unclear how this biomarker develops after liver transplantation and how valid its predictions are for post-operative infections.

Therefore, patients scheduled for liver transplantation will be included in the trial. AGRA measurements before and after the transplant (1, 7, 90 days after the end of antibiotic treatment) will be performed. Additionally outcome data regarding severe infections are collected for one year before and after transplantation. The respective organ donors are included as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-80 years
* Listed for liver transplantation (for recipients)
* Liver recipient is included in the study (for donors)
* Informed consent

Exclusion Criteria:

* Antibiotic therapy with substances active against E. coli at the scheduled blood sampling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for liver transplantation at the University Hospital in Graz, Austria for any reason will be included in the study. The respective donors will serve as a control cohort.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of Acellular growth retardation ability (AGRA) | change from transplantation to 90 days after the end of prophylactic antibiotic treatment after the transplantation
  Functional biomarker for the state of the humoral immune system

SECONDARY OUTCOMES:
Infections | 1 year after transplantation
  Occurrence of severe infections
Infections | 1 year before transplantation
  Occurrence of severe infections
Complications | during hospital stay
  Occurrence of transplantation-related complications
C reactive protein | change from transplantation to 90 days after the end of prophylactic antibiotic treatment after the transplantation
  routine biomarker for infections
Liver function | before transplantation
  State of the donated liver, including results of a possible liver biopsy prior to transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Geraz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided